CLINICAL TRIAL: NCT05522595
Title: Evaluation of the Performance and Safety of the S360 Medical Device Software.
Brief Title: Performance and Safety Evaluation of the S360 Medical Device Software.
Acronym: ArgoS360
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sierra Neurovision (Industry)
Collaborators: Institut des Sciences de la Vision (Unknown); CEISO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S360 IC-01
Record Dates: First submitted 2022-08-23; First posted 2022-08-31 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-08

CONDITIONS: Binocular Vision Disorder; Binocular Eye Movement Disorder; Ocular Motion; Disorder
Keywords: Eye tracker; Orthoptics analysis; Neuro-visuo-motor analysis; Eye movement
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care arm (Experimental): The patient is his own comparator. During the intervention, the eyes movements measurements will be performed using the standard of care and the medical device S360.
  Interventions: Device: S360

INTERVENTIONS:
Device: S360 — In the first part of the intervention, after the CISS questionnaire completion by the patient, participant's eyes movements measurement will be performed using the reference procedure (standard of care).
  A first diagnosis is established according to the interpretation of the results by a first evaluator.
  In the second part of the intervention, the participant's eyes movements will be measured using the medical device S360.
  A second diagnosis is established according to the interpretation of the software's displayed data by a second evaluator.

SUMMARY:
The aim of this interventional, cross-sectional study is to evaluate the performance and the safety of the medical device software S360. This clinical investigation is performed in order to demonstrate the conformity of the medical device, when operating under the normal conditions of its intended use, in accordance with the General Safety and Performance Requirements pertaining to clinical evaluation of the device regarding the Medical Device Regulation (MDR) 2017/745 (EU).

DETAILED DESCRIPTION:
Background:

Accurate detection and interpretation of eye movement abnormalities often guides differential diagnosis and discussions on prognosis. Therefore, adequate diagnosis permits to direct treatment of disabling visual symptoms and signs. A comprehensive clinical eye movement examination is high yield from a diagnostic standpoint; however, skilful recording and quantification of eye movements can increase detection of subclinical deficits, confirm clinical suspicions, guide therapeutics, and generate expansive research opportunities.

Recently, many technologies, allowing objective measurements, have been developed. The most commonly used eye movement measurement technique is the high frequency video camera (Eye tracker).

In this context, SIERRA NEUROVISION has developed the S360, a medical device software using the infrared video-oculography technology. It is intended to collect data for orthoptics and neuro-visuo-motor analysis. It records the patient's eye movements, displays the patient's scoring next to normative values retrieved from literature and widely used in the current practice.

Design:

The study is cross-sectional, interventional, open label, single-arm, comparative and single-center study.

This study is a pre-marketing, confirmatory research which is performed in order to evaluate the performance and the safety of S360 MDSW compared to the standard of care procedure.

Intervention:

As the current study is cross-sectional, no follow-up visits related to the study are planned. All study procedures will be carried out during the inclusion visit which will take place during the patient's medical visit as part as his/her standard of care.

The study will be conducted in two parts:

Part 1 : standard of care measurements.

* CISS (Screening for convergence insufficiency) questionnaire completion
* Eye movements measurements using the standard tools used by the orthoptist (a prism bar, a penlight and a video projector, etc).

A first diagnosis based on the interpretation of the results provided by the standard of care measurements will be established by a first evaluator (orthoptist).

Part 2: S360 measurements

- Eye movements measurements using the medical device software S360. A second diagnosis based on the interpretation of the outcomes provided by the MDSW S360 will be established by a second evaluator (orthoptist).

The two measurements procedures are performed in two different examination rooms by two different operators. The diagnoses are established by two different investigators (orthoptist).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 6 years old requiring an orthoptic or neuro-visual assessment in order to assess the effectiveness of oculomotor skills;
* Both gender; male and female
* Symptomatic or non-symptomatic patient;
* Affiliated person or beneficiary of a social security scheme,
* Free, informed and written consent signed by the participant and the investigator for adults or by parents/legal representative for patients aged from 6 to 17years old

Exclusion Criteria:

* Visual acuity below 5/10 not improvable
* Patient with a head injury;
* Patient with ocular injury;
* Patient with diagnosed serious pathologies that may interfere with the study measurements;
* Patient with medical treatment that may interfere with the study
* Patient with hypersensitivity to electronic devices;
* Non-cooperative patient (e.g. restless patient);
* Non-French speaker patient;
* Patient unable to understand study procedures;
* Subject who has forfeited their freedom by administrative or legal award, or is under guardianship or under limited judicial protection;
* Patient refusing to participate in the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (Se) and specificity (Sp) | Day 0
  Sensitivity (Se) and specificity (Sp) of performed diagnosis using recorded data from the S360 versus performed diagnosis with standard measurement

SECONDARY OUTCOMES:
Accuracy of the S360's measured data | Day 0
  Error rate calculation of the S360's measured data
Repeatability of the S360's measured data | Day 0
  Coefficient of variation calculation of the S360's measured data
Reproducibility of the S360's measured data | Day 0
  The reproducibility coefficient of the S360's measured data
Evaluation of the usefulness of the MDSW S360 in the current practice | Day 0
  Rate of positive feedback estimation
Validation of the technical functionalities of the MDSW S360 | Day 0
  Calculation of the :
  * Rate of successful outcomes transmission
  * Rate of successful display of outcomes measurement
  * Rate of successful report generation
  * Rate of successful report transmission
Safety : Adverse events | Day 0
  Incidence of the medical device's related-adverse events estimation
Operator's comfort of using the medical device S360 | Day 0
  Operator's comfort of using the medical device and the headset survey Comfort level will be expressed by the rate of satisfaction: Higher rate means a better Comfort
Comparison of the duration of the two procedure | Day 0
  Average duration of the two procedures (S360 vs Standard of care)
Patient satisfaction | Day 0
  Patient's satisfaction level by using a satisfaction survey Satisfaction level will be expressed by the rate of satisfaction: Higher rate means a better satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Maleysson, Principal Investigator — Institut des Sciences de la Vision
Locations (1):
- Institut des Sciences de la Vision, Saint-Etienne, France